CLINICAL TRIAL: NCT01971619
Title: Association of Vitamin D, Parathyroid Hormone and Fibroblast Growth Factor-23 With Infarction-related Arrhythmia in Patients With Acute Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2013-0424
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma blood sample (5ml)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SACS cohort: patients with acute myocardial infarction at Severance hospital

SUMMARY:
To investigate the effect of vitamin D deficiency on the development of arrhythmia in patients with acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* age ≥20 years
* diagnosed with acute myocardial infarction (confirmed by cardiac enzyme and EKG)
* subjects who agreed with informed consent

Exclusion Criteria:

* previous history of arrhythmia before onset of acute myocardial infarction
* currently taking anti-arrhythmic drugs
* severe condition of comorbid diseases that can cause more serious effects on patients than acute myocardial infarction does (e.g., cancer, cerebrovascular diseases, acute bleeding etc.)

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute myocardial infarction
Sampling Method: Probability Sample
Enrollment: 510 (Estimated)
Dates: Start 2013-08; Primary Completion 2013-10 (Actual); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Events of acute myocardial infarction-associated arrhythmia | first 48 hours after onset of acute myocardial infarction
  incidence of acute myocardial infarction-associated arrhythmia types of arrhythmia, duration of arrhythmia, persistence of arrhythmia

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Rienstra M, Cheng S, Larson MG, McCabe EL, Booth SL, Jacques PF, Lubitz SA, Yin X, Levy D, Magnani JW, Ellinor PT, Benjamin EJ, Wang TJ. Vitamin D status is not related to development of atrial fibrillation in the community. Am Heart J. 2011 Sep;162(3):538-41. doi: 10.1016/j.ahj.2011.06.013. Epub 2011 Aug 11. PMID 21884873